CLINICAL TRIAL: NCT06930352
Title: Frontline Ziftomenib in NPM1-Mutated or KMT2A-Rearranged Acute Myeloid Leukemia in Patients Not Eligible for Intensive Induction or Other Therapy
Brief Title: Ziftomenib for the Treatment of Patients With NPM1 Mutated or KMT2A Rearranged Acute Myeloid Leukemia Not Eligible for Standard Therapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Uma Borate (Other)
Collaborators: Kura Oncology (Unknown)
Responsible Party: Sponsor-Investigator, Uma Borate, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-24309; NCI-2025-02414 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; Cytarabine; Hydroxyurea; Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (ziftomenib) (Experimental): Patients receive ziftomenib PO QD on days 1-28 of each cycle. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients may also undergo cytoreduction therapy with hydroxyurea up to end of cycle 1, cytarabine within 7 days of starting treatment, or leukapheresis within 7 days of treatment to reduce white blood cell count to =< 10,000/uL. Additionally, patients undergo ECHO or MUGA at screening and bone marrow biopsy and/or aspiration and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Cytarabine; Procedure: Echocardiography Test; Drug: Hydroxyurea; Procedure: Leukapheresis; Procedure: Multigated Acquisition Scan; Other: Questionnaire Administration; Drug: Ziftomenib

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow biopsy and/or aspiration
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy and/or aspiration
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Cytarabine — Given cytarabine
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Hydroxyurea — Given hydroxyurea
  Other Names: Droxia; Hydrea; Hydroxycarbamide; Litalir; Onco-Carbide; Oncocarbide; Oxeron; SQ 1089; SQ-1089; Syrea; WR 83799
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocyte Adsorptive Apheresis; Leukocytopheresis; Therapeutic Leukopheresis; White Blood Cell Reduction Apheresis
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Other: Questionnaire Administration — Ancillary studies
Drug: Ziftomenib — Given PO
  Other Names: KO 539; KO-539; KO539; Menin-KMT2A Inhibitor KO 539; Menin-Mixed Lineage Leukemia Protein-Protein Interaction Inhibitor KO 539; Menin-MLL Inhibitor KO-539; Menin-MLL Interaction Inhibitor KO 539

SUMMARY:
This phase II trial tests how well ziftomenib works in treating patients with NPM1 mutated or KMT2A rearranged acute myeloid leukemia (AML) and are not eligible to receive standard therapy. AML is often due to genetic changes in the cancer cells, including mutations in the NPM1 gene and rearrangements involving the KMT2A gene. These mutations result in activation of the menin pathway. Menin is a type of protein in the body that helps to regulate some of the naturally occurring processes in the body, but can also be involved in some types of cancers. Ziftomenib blocks this menin pathway and may prevent the cancer cells from continuing to grow. Giving ziftomenib may kill more cancer cells in patients with NPM1 mutated or KMT2A rearranged AML that are not eligible to receive standard therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the efficacy of ziftomenib in treatment-naïve patients with KMT2A-rearranged (r) and NPM1-mutated (m) AML who are not candidates for standard therapy, with primary endpoint of complete remission (CR) + CR/response with hematologic improvement (CRh), assessed after 6 cycles of treatment using the best response achieved in that time.

SECONDARY OBJECTIVES:

I. To determine rates of transfusion independence for 8- and 16-week periods. II. To determine response including CR, composite CR (CRc) (CR + CRh + CR with incomplete blood count recovery [CRi] + CR with incomplete platelet recovery [CRp]), proportion of patients achieving CRc with negative measurable residual disease (MRD), overall response rate (ORR) (CRc + partial response [PR] + morphologic leukemia free state [MLFS]).

III. To determine duration of response (DOR). IV. To determine overall survival (OS), and event free survival (EFS) at 24 months.

V. To evaluate if ziftomenib treatment improves quality of life using the Patient Reported Outcomes Measurement Information System (PROMIS)-29+2 version (v) 2.1 questionnaire.

VI. To assess safety in this patient population by determining the number of patients experiencing adverse events/serious adverse events.

EXPLORATORY OBJECTIVES:

I. To assess efficacy in patients with mutations thought to be sensitive to menin inhibition, other than KMT2A rearrangements and NPM1 mutations.

II. To perform measurable residual disease (MRD) monitoring via liquid biopsy to monitor clonal dynamics during treatment.

III. To assess the clonal, biochemical and differentiation changes in AML cells during treatment with menin inhibition using flow cytometry, cytogenetics and serial next generation sequencing on bone marrow specimens before and during treatment to assess for potential resistance mutations or clonal evolution that may be predictors of relapse.

OUTLINE:

Patients receive ziftomenib orally (PO) once daily (QD) on days 1-28 of each cycle. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients may also undergo cytoreduction therapy with hydroxyurea up to end of cycle 1, cytarabine within 7 days of starting treatment, or leukapheresis within 7 days of treatment to reduce white blood cell count to =< 10,000/uL. Additionally, patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) at screening and bone marrow biopsy and/or aspiration and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 6 months for up to 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study
* Morphologically confirmed diagnosis of the following based on 2022 World Health Organization (WHO) Classification:

  * Treatment-naïve acute myeloid leukemia
  * KMT2A rearrangement (defined as KMT2A translocations) OR NPM1 mutation (defined as NPM1 mutation resulting in cytoplasmic localization, or NPM1c) OR other mutations that have been shown to exhibit sensitivity to menin inhibition. Mutation status will be known from initial diagnosis using standard of care testing, which can be performed locally
* Patients ineligible or unwilling to receive standard of care induction therapy, such as 7+3, hypomethylating agent, venetoclax, or other standard of care (SOC) regimens with ineligibility defined by the following:

  * ≥ 75 years of age with both of the following;

    * Subject must have adequate renal function as demonstrated by a creatinine clearance ≥ 30 mL/min; calculated by the Cockcroft Gault formula or measured by 24-hours urine collection
    * Subject must have adequate liver function as demonstrated by aspartate aminotransferase (AST) ≤ 3.0 x upper limit of normal (ULN) and alanine aminotransferase (ALT) ≤ 3.0 x ULN (unless considered due to leukemic organ involvement) OR
  * ≥ 18 to 74 years of age with at least one of the following co-morbidities:

    * Eastern Cooperative Oncology Group (ECOG) performance status of 2 or 3;
    * Cardiac history of congestive heart failure (CHF) requiring treatment or ejection fraction ≤ 50% or chronic stable angina;
    * Diffusion capacity of the lung for carbon monoxide (DLCO) ≤ 65% or forced expiratory volume in 1 second (FEV1) ≤ 65%;
    * Creatinine clearance ≥ 30 mL/min to < 45 ml/min;
    * Moderate hepatic impairment with total bilirubin > 1.5 to ≤ 3.0 x ULN;
    * Venous thromboembolism benefitting from prolonged anticoagulation or presence of prosthetic heart valve or any indication for therapeutic anticoagulation with a single agent
    * Prior history of severe infection requiring hospitalization with risk of recurrence with subsequent immunosuppression
    * Any other comorbidity that the physician judges to be incompatible with standard frontline therapy must be reviewed and approved by the study team before study enrollment
* Peripheral white blood cell (WBC) counts ≤ 10,000/uL. Patients may receive hydroxyurea, cytarabine, or leukapheresis to control and maintain white blood cell count until the end of cycle 1
* Women of childbearing potential must be willing to use a highly effective method of contraception throughout the study and for at least 180 days after the last dose of study treatment
* Non-sterile male patients must agree to use a highly effective method of contraception with partner(s) throughout the study and for at least 90 days after the last dose of study treatment

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia
* Diagnosis of chronic myelogenous leukemia in blast crisis
* Clinically active central nervous system (CNS) leukemia
* Prior treatment for AML except for hydroxyurea and/or cytarabine used for control of leukocytosis
* Treatment with concomitant drugs that are strong inhibitors or inducers of cytochrome P450-isozyme 3A4 (CYP3A4) with the exception of antibiotics, antifungals, and antivirals that are used as standard of care or to prevent or treat infections and other such drugs that are considered absolutely essential for the care of the patient
* Detectable viral load for human immunodeficiency virus, hepatitis C, or hepatitis B surface antigen indicative of active infection. Patients with controlled disease will not be excluded from study enrollment
* Pre-existing disorder predisposing the patient to a serious or life-threatening infection (e.g. cystic fibrosis, congenital or acquired immunodeficiency, bleeding disorder, or cytopenias not related to AML)
* Active uncontrolled acute or chronic systemic fungal, bacterial, viral, or other infection
* Mean Fridericia's formula-corrected QT interval (QTcF) > 480 ms on triplicate electrocardiogram (ECG)
* Any psychiatric illness that prevents patient from informed consent process
* Women who are pregnant or lactating. All female patients with reproductive potential must have a negative serum pregnancy test within 72 hours prior to starting treatment
* Participants requiring dual antiplatelet therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission (CR) plus CR/response with hematologic improvement | After 6 cycles of treatment (cycle length = 28 days)
  Will be assessed after 6 cycles of treatment using the best response achieved in that time. Will be calculated in each arm for the efficacy analysis population and reported along with two-sided 95% exact binomial confidence limits, in a modified intent-to-treat analysis.

SECONDARY OUTCOMES:
Rate of transfusion independence | Up to 24 months
  Transfusion independence is defined as the proportion of subjects without transfusions during any consecutive 8 weeks (56 days) starting from Study Day 1 and has correlated with palliative benefits in patients with AML [19]. The major criteria for judging response will include physical examination and laboratory evaluation.
CR rate | Up to 24 months
  Will also be calculated in the primary efficacy analysis cohort along with 95% exact binomial confidence intervals.
Composite CR (CRc) rate | Up to 24 months
  Will also be calculated in the primary efficacy analysis cohort along with 95% exact binomial confidence intervals.
CRc with negative measurable residual disease | Up to 24 months
  Will also be calculated in the primary efficacy analysis cohort along with 95% exact binomial confidence intervals.
Overall response rate | Up to 24 months
  Will also be calculated in the primary efficacy analysis cohort along with 95% exact binomial confidence intervals.
Duration of response | From the date first achieved response to the date of progression or relapse or death, whichever occurs first, assessed up to 24 months
  Will be estimated using the method of Kaplan-Meier and calculated in the primary efficacy analysis.
Overall survival | From date of treatment start to death due to all causes, assessed up to 24 months
  Will be estimated using the method of Kaplan-Meier and calculated in the primary efficacy analysis.
Event free survival | From initiation of study treatment to the date of confirmed progressive disease, confirmed morphological relapse, treatment failure after 6 cycles of study treatment (cycle length = 28 days) or death from any cause, assessed up to 24 months
  Will be estimated using the method of Kaplan-Meier and calculated in the primary efficacy analysis.
Changes in quality of life | Day 1 of each cycle up to completion of treatment (cycle length = 28 days)
  Will be measured using Patient Reported Outcomes Measurement Information System (PROMIS) 29 +2 version (v) 2.1 and Patient Reported Outcomes (PRO) Common Terminology Criteria for Adverse Events (CTCAE). The raw sum will be calculated and converted to the standardized T score. Descriptive statistics will be used to present the PROMIS and PRO-CTCAE scores at each time point, and we will also use graphical display to visualize the change in quality of life over time. Wilcoxon signed rank test will be used to test if the change over time is statistically significant. To further quantify the change over time, linear mixed model will be fit for PROMIS score and PRO-CTCAE score, and if the sample size allows, the model will control for important clinical covariates as well.
Incidence of adverse events (AEs) | Up to 30 days after last dose of study treatment
  AEs will be graded according to CTCAE v 5.0. The toxicity data captured will include type, frequency, grade, severity, timing of onset, duration, and relationship to study drug. Frequency tables will be used to summarize the AE data, where the number of patients with different types of AE will be tabulated by toxicity grade, counting only the highest grade of a certain type of AE occurred to the same patient. All adverse events regardless of attribution as well as those treatment-related AEs will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Uma M Borate, MBBS, MD, MSc, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu